CLINICAL TRIAL: NCT03851419
Title: The Burden of (Neuro)Cysticercosis Among People Living With HIV Compared With HIV-negative Individuals in the Rural Southern Highlands in Tanzania
Brief Title: The Burden of (Neuro)Cysticercosis Among People Living With HIV in Rural Tanzania
Acronym: CYSTINET_Tz
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Kilimanjaro Clinical Research Institute (Other); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CYSTINET-Africa Tz II
Record Dates: First submitted 2019-02-04; First posted 2019-02-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Neurocysticercosis; HIV/AIDS
MeSH Terms: conditions — Neurocysticercosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People living with HIV: People living with HIV (ART naive or on ART)
  Interventions: Diagnostic Test: Diagnosis of (Neuro)cysticercosis
- People not infected with HIV: HIV-negative people. Each participant is matched for age, sex and location to a study participant living with HIV
  Interventions: Diagnostic Test: Diagnosis of (Neuro)cysticercosis

INTERVENTIONS:
Diagnostic Test: Diagnosis of (Neuro)cysticercosis — * Serological tests for cysticercosis
  * Neurological examination and cerebral CT scan for the diagnosis of neurocysticercosis
  * Stool testing for T. solium

SUMMARY:
This study aims to compare the burden of neurocysticercosis among people living with HIV to people not infected with HIV.

DETAILED DESCRIPTION:
People living with HIV and matched HIV negative controls will be tested serologically for cysticercosis, examined neurologically and will undergo CT scanning to determine the prevalence and presentation of NCC.

Furthermore, the immune system response in HIV patients with Taenia solium neurocysticercosis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who consent to participate in the study and testing.
* Patients of age 14 years and above
* Patient living inside the study catchment area
* HIV-positive patients
* Patient suspected of taeniasis or cysticercosis/neurocysticercosis

Exclusion Criteria:

* Patients with opportunistic infections.
* Study participants taking anthelminthic drugs PZQ and ALB or have received them within the previous 12 months.
* Pregnant women
* Patients that are seriously ill.
* Patients with epilepsy and other mental disorders that impair thoughts and emotions such as psychosis.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1000 patients from HIV clinics will be recruited at the study sites in Mbeya and Iringa region. For each HIV-positive patient an HIV-negative control matched by age, sex and location will be included.
Sampling Method: Non-Probability Sample
Enrollment: 2584 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of cysticercosis | Single assessment at inclusion into study (serological testing)
  Prevalence of cysticercosis among people living with HIV and matched HIV-negative individuals in rural Tanzania where pig farming is common
Prevalence of neurocysticercosis | Single assessment through cerebral CT scan at inclusion into study
  Prevalence of neurocysticercosis among people living with HIV and matched HIV-negative individuals in rural Tanzania where pig farming is common

SECONDARY OUTCOMES:
Th1 cytokines among neurocysticercosis patients | One time assessment through immunological testing at inclusion into study
  To compare the specific peripheral immune response against T. solium neurocysticercosis between symptomatic and asymptomatic patients measured by concentration of Th1 cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard J Ngowi, MD, PhD, Principal Investigator — National Institute for Medical Research
Locations (1):
- National Institute of Medical Research, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided